CLINICAL TRIAL: NCT07107620
Title: Investigation of Dual Task Performance of Individuals With Type 2 Diabetes Mellitus
Brief Title: Dual Task Performance and Type II Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Abdulkadir Ertürk, Principal Investigator, Kahramanmaras Sutcu Imam University
Other Study IDs: KSÜKADİRERTÜRK1
Record Dates: First submitted 2025-06-28; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Type II Diabetes Mellitus; Dual Task Cost
Keywords: Type II Diabetes Mellitus; Dual-task; Cognition
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type II diabetes mellitus group: Dual task tests were applied to the group with type 2 diabetes mellitus
  Interventions: Diagnostic Test: one task; Diagnostic Test: dual task
- Healthy group: Dual task tests were administered to the healthy group
  Interventions: Diagnostic Test: one task; Diagnostic Test: dual task

INTERVENTIONS:
Diagnostic Test: one task — Single task tests consist of measuring walking times with normal walking (easy), walking with a 50% reduction in the base of support measured between the medial malleoli (medium difficulty) and tandem walking (difficult) tasks while applying the 10 meter walk test and time up go tests.
Diagnostic Test: dual task — Dual task consists of single task plus tests of carrying glasses of water or counting backwards from a given number.

SUMMARY:
The aim of this study is to compare the dual task performances of individuals with and without type 2 diabetes. Thus, it will be concluded whether having type 2 diabetes affects dual task performance.

DETAILED DESCRIPTION:
In our daily lives, we often have to juggle many tasks simultaneously. Performing two tasks simultaneously is called dual-tasking. The ability to perform two tasks simultaneously is called dual-tasking performance. Dual-tasking performance can decrease in individuals with diabetes due to complications of diabetes. This study compared the dual-tasking performance of individuals with type 2 diabetes and healthy individuals using dual-tasking tests categorized as easy, medium, and difficult.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type II DM (for the Type II diabetes group)
* Being 50 years old or older
* Being a native Turkish speaker

Exclusion Criteria:

* Not being able to read and write,

  * Having communication problems,
  * Having a score below 24 points on the Standardized Mini-Mental Test,
  * Having one of the neurological diseases that will affect the study such as Parkinson's, stroke, etc.,
  * Having upper and/or lower extremity surgery in the last year or having a surgical history that will affect walking,
  * Having retinopathy, foot ulcers, and severe sensory impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have had diabetes for at least 1 year and are over 50 years of age and their matched healthy controls constitute the study sample.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
10 meter walk test | one day
  The dual task cost was calculated to measure dual task performance by applying the 10-meter walking test as single and dual tasks.
  This cost will be calculated as follows:
  (Dual task performance-single task performance)/ single task performance x100
time up go test | one day
  The dual task cost was calculated to measure dual task performance by applying the time up go test as single and dual tasks. This cost will be calculated as follows: (Dual task performance-single task performance)/ single task performance x100

SECONDARY OUTCOMES:
Stroop test | one day
  There are 5 sections in this test. Section 1 includes reading black text, section 2 includes reading colored words related to color names, section 3 includes saying the color of shapes, section 4 includes saying the color of words that are not color names, and section 5 includes saying the color of colored words that are color names. Individuals are asked to read from left to right as fast as possible. The time taken is recorded in seconds.
Dual task survey | one day
  It is a test that questions the difficulties experienced by individuals during dual-task activities in daily life activities. The survey consists of 10 questions. The short duration of the survey is an advantage. The survey, which consists of 5 answers, is scored between 0 and 4. A score of ''4'' indicates that difficulties are experienced very often, ''0'' indicates that there is no difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Suat EREL, professor, Study Director — Pamukkale University Faculty of Health Sciences
Locations (1):
- Pamukkale University hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No